CLINICAL TRIAL: NCT02347072
Title: A Randomized, Phase IIIb, Three-period, Three-treatment, Double-blind, Multi-center, Crossover Study to Evaluate the 24-hour Lung Function Profile in Subjects With Moderate to Very Severe COPD After 4 Weeks of Treatment With PT003, Open-Label Spiriva® Respimat® (Tiotropium Bromide) as an Active Control, and Placebo
Brief Title: 24-hour Lung Function in Subjects With Moderate to Very Severe COPD After Treatment With PT003, Open-Label Spiriva® Respimat® as an Active Control, and Placebo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PT003011-00
Record Dates: First submitted 2015-01-21; First posted 2015-01-27 (Estimated); Results first posted 2017-04-19 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2017-03

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Glycopyrrolate; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- GFF MDI (PT003) (Experimental): Glycopyrronium and Formoterol Fumarate Inhalation Aerosol; PT003, Glycopyrronium and Formoterol Fumarate Metered Dose Inhaler (GFF MDI)
  Interventions: Drug: GFF MDI (PT003)
- Placebo MDI (Placebo Comparator): Placebo Metered Dose Inhaler (MDI) for Glycopyrronium and Formoterol Fumarate Inhalation Aerosol
  Interventions: Drug: Placebo MDI
- Spiriva® Respimat® (Tiotropium Bromide) (Active Comparator): Tiotropium Bromide Inhalation Solution; Spiriva® Respimat® (Spiriva)
  Interventions: Drug: Spiriva® Respimat® (Tiotropium Bromide)

INTERVENTIONS:
Drug: GFF MDI (PT003)
  Other Names: Glycopyrronium and Formoterol Fumarate Inhalation Aerosol; PT003, Glycopyrronium and Formoterol Fumarate Metered Dose Inhaler (GFF MDI)
  Arms: GFF MDI (PT003)
Drug: Placebo MDI
  Other Names: Placebo Metered Dose Inhaler (MDI) for Glycopyrronium and Formoterol Fumarate Inhalation Aerosol
  Arms: Placebo MDI
Drug: Spiriva® Respimat® (Tiotropium Bromide) — Tiotropium Bromide Inhalation Solution; Spiriva® Respimat® (Spiriva)
  Arms: Spiriva® Respimat® (Tiotropium Bromide)

SUMMARY:
Randomized, Phase IIIb, Three-period, Three-treatment, Double-blind, Multi-center, Crossover Study to Evaluate the 24-hour Lung Function Profile in Subjects with Moderate to Very Severe COPD after 4 Weeks of Treatment with PT003, Open-Label Spiriva® Respimat® (Tiotropium Bromide) as an Active Control, and Placebo.

ELIGIBILITY:
Inclusion Criteria:

* At least 40 years of age and no older than 80 at Screening
* Women of non-child bearing potential or negative serum pregnancy test at Screening, and agrees to acceptable contraceptive methods used consistently and correctly Screening until 14 days after final visit.
* Subjects with an established clinical history of COPD as defined by the American Thoracic Society (ATS)/European Respiratory Society (ERS)
* Current or former smokers with a history of at least 10 pack-years of cigarette smoking
* Pre- and post-bronchodilator FEV1/FVC ratio of <0.70
* Post-bronchodilator FEV1 must be <80% predicted normal value, calculated using NHANES III reference equations, and the measured FEV1 must also be ≥750 mL if FEV1 <30% of predicted normal value.

Exclusion Criteria:

* Significant diseases other than COPD, i.e., disease or condition which, in the opinion of the Investigator, may put the subject at risk because of participation in the study or may influence either the results of the study or the subject's ability to participate in the study.
* Women who are pregnant or lactating.
* Subjects, who in the opinion of the Investigator, have a current diagnosis of asthma.
* Subjects who have been hospitalized due to poorly controlled COPD within 3 months prior to Screening or during the Screening Period.
* Subjects who have poorly controlled COPD, defined as acute worsening of COPD that requires treatment with oral corticosteroids or antibiotics within 6 weeks prior to Screening or during the Screening Period.
* Subjects who have clinically significant uncontrolled hypertension.
* Subjects who have cancer that has not been in complete remission for at least five years.
* Subjects with abnormal liver function tests defined as AST, ALT, or total bilirubin ≥1.5 times upper limit of normal at Screening and on repeat testing.
* Subjects with a diagnosis of angle closure glaucoma will be excluded, regardless of whether or not they have been treated. Subjects with a diagnosis of open angle glaucoma who have intraocular pressure controlled with medication(s) are eligible.
* Subjects with symptomatic prostatic hypertrophy that is clinically significant in the opinion of the Investigator. Subjects with a trans-urethral resection of prostate (TURP) or full resection of the prostate within 6 months prior to Screening are excluded from the study.
* Subjects with bladder neck obstruction or urinary retention that is clinically significant in the opinion of the Investigator.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2015-08-01 (Actual); Study Completion 2016-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colin Reisner, MD, Study Chair — Pearl Therapeutics

REFERENCES:
- [Derived] Reisner C, Gottschlich G, Fakih F, Koser A, Krainson J, Delacruz L, Arora S, Feldman G, Pudi K, Siddiqui S, Orevillo C, Maes A, St Rose E, Martin U. 24-h bronchodilation and inspiratory capacity improvements with glycopyrrolate/formoterol fumarate via co-suspension delivery technology in COPD. Respir Res. 2017 Aug 18;18(1):157. doi: 10.1186/s12931-017-0636-4. PMID 28821260

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 10 sites in the US from February 2015 to August 2015. The study was anticipated to run for approximately 9 months but not expected to exceed 12 months.
Pre-assignment Details: Study to assess the efficacy and safety of GFF MDI 14.4/9.6µg relative to either Placebo MDI or Spiriva Respimat 5µg. Subjects were randomized into 1 of 6 treatment sequences, and all treatment sequences included all 3 treatments. By-treatment sequence tabulations of the data were not pre-specified.
Groups:
- Overall Study: All Subjects Randomized
Period: Overall Study
Arm/Group | Overall Study
Started | 80
GFF MDI 14.4/9.6 µg | 75
Placebo MDI | 72
Spiriva Respimat 5 µg | 73
Completed | 62
Not Completed | 18
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 6
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 2
Not completed — Protocol Violation | 1
Not completed — Disc due to Protocol-specified Criteria | 6

BASELINE CHARACTERISTICS:
Population: MITT population was a subset of the ITT Population including subjects who received treatment and had post treatment efficacy data from at least 2 treatment periods and this population is used for baseline characteristics. Participant Flow includes all patients randomized, regardless of treatment received.
Arm/Group | All Subjects
Number analyzed (Participants) | 75
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.8 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 27

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Area Under the Curve (AUC) 0-24
Description: Normalized Forced Expiratory Volume in 1 second (FEV1) Area Under the Curve (AUC) 0-24
Time Frame: Pre dose, 15 and 30 minutes, 1, 2, 4, 8, 12, 12.25, 12.5, 13, 14, 16, 22, and 24 hours post the morning dose on Day 29
Population: Subjects in the Modified Intent to Treat (MITT) Population who had a sufficient number of post dose FEV1 measurements
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Groups:
- GFF MDI: Glycopyrronium Formoterol GFF Metered Dose Inhaler MDI 14.4/9.6µg
- Spiriva Respimat: Spiriva Respimat 5μg
- Placebo: Placebo MDI
Arm/Group | GFF MDI | Spiriva Respimat | Placebo
Number analyzed (Participants) | 65 | 67 | 65
Liters | 0.192 [0.141 to 0.243] | 0.112 [0.061 to 0.162] | -0.072 [-0.123 to -0.022]

2. Secondary Outcome: FEV1 AUC12-24
Description: Normalized FEV1 AUC12-24
Time Frame: Pre dose, 15 and 30 minutes, 1, 2, 4, 8, and 12 hours post the evening dose on Day 29
Population: Subjects in the MITT Population who had a sufficient number of post dose FEV1 measurements
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | GFF MDI | Spiriva Respimat | Placebo
Number analyzed (Participants) | 65 | 67 | 65
Liters | 0.159 [0.104 to 0.214] | 0.039 [-0.015 to 0.094] | -0.118 [-0.173 to -0.063]

3. Secondary Outcome: FEV1 AUC0-12
Description: Normalized FEV1 AUC0-12
Time Frame: Pre dose, 15 and 30 minutes, 1, 2, 4, 8, and 12 hours post the morning dose on Day 29
Population: Subjects in the MITT Population who had a sufficient number of post dose FEV1 measurements
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | GFF MDI | Spiriva Respimat | Placebo
Number analyzed (Participants) | 67 | 68 | 66
Liters | 0.226 [0.175 to 0.276] | 0.178 [0.127 to 0.228] | -0.026 [-0.077 to 0.025]

4. Secondary Outcome: Peak Change From Baseline in FEV1 Evening
Description: Peak Change From Baseline in FEV1 Evening
Time Frame: Baseline and Day 29
Population: MITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | GFF MDI | Spiriva Respimat | Placebo
Number analyzed (Participants) | 65 | 67 | 65
Liters | 0.395 [0.334 to 0.456] | 0.230 [0.170 to 0.291] | 0.058 [-0.003 to 0.119]

5. Secondary Outcome: Peak Change From Baseline in FEV1 Morning
Description: Peak Change From Baseline in FEV1 Morning
Time Frame: Baseline and Day 29
Population: Subjects in the MITT Population who had a sufficient number of post dose FEV1 measurements
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | GFF MDI | Spiriva Respimat | Placebo
Number analyzed (Participants) | 67 | 68 | 67
Liters | 0.406 [0.351 to 0.462] | 0.325 [0.270 to 0.381] | 0.129 [0.073 to 0.185]

6. Secondary Outcome: Morning Pre-Dose Trough FEV1 on Day 29
Description: Morning Pre-Dose Trough FEV1 on Day 29
Time Frame: Day 29
Population: Subjects in the MITT Population who had a sufficient number of post dose FEV1 measurements
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | GFF MDI | Spiriva Respimat | Placebo
Number analyzed (Participants) | 67 | 68 | 66
Liters | 0.140 [0.095 to 0.185] | 0.097 [0.053 to 0.142] | -0.020 [-0.066 to 0.025]

7. Secondary Outcome: Morning Pre-Dose Trough FEV1 on Day 30
Description: Morning Pre-Dose Trough FEV1 on Day 30
Time Frame: Day 30
Population: Subjects in the MITT Population who had a sufficient number of post dose FEV1 measurements
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | GFF MDI | Spiriva Respimat | Placebo
Number analyzed (Participants) | 66 | 66 | 66
Liters | 0.129 [0.073 to 0.185] | 0.072 [0.015 to 0.128] | -0.073 [-0.130 to -0.017]

8. Secondary Outcome: Peak Change From Baseline in IC (Inspiratory Capacity) Evening
Description: Peak Change From Baseline in IC Evening
Time Frame: Baseline and Day 29
Population: Subjects in the MITT Population who had a sufficient number of post dose FEV1 measurements
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | GFF MDI | Spiriva Respimat | Placebo
Number analyzed (Participants) | 62 | 67 | 63
Liters | 0.421 [0.343 to 0.498] | 0.297 [0.221 to 0.372] | 0.109 [0.032 to 0.186]

9. Secondary Outcome: Peak Change From Baseline in IC Morning
Description: Peak Change From Baseline in IC Morning
Time Frame: Baseline and Day 29
Population: Subjects in the MITT Population who had a sufficient number of post dose FEV1 measurements
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | GFF MDI | Spiriva Respimat | Placebo
Number analyzed (Participants) | 67 | 66 | 65
Liters | 0.454 [0.388 to 0.520] | 0.374 [0.307 to 0.440] | 0.206 [0.139 to 0.273]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the subject signed consent up to the follow-up phone call 7-14 days after last dose of study drug.
Description: The Safety Population was defined as all subjects who were randomized to treatment and received at least one dose of study treatment. Serious adverse events collected from time of consent up to 14 days after last dose of study drug.
Arm/Group | GFF MDI | Spiriva Respimat | Placebo
Serious Adverse Events (participants affected / at risk) | 2/75 | 2/73 | 2/72
Other Adverse Events (participants affected / at risk) | 5/75 | 5/73 | 6/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GFF MDI (N=75) | Spiriva Respimat (N=73) | Placebo (N=72)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GFF MDI (N=75) | Spiriva Respimat (N=73) | Placebo (N=72)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Tremor (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Drafts of any and all publications or presentations of this study must be submitted at least 30 days prior to submission for publication or presentation to Pearl Therapeutics for review, approval, and to ensure consistency. Pearl Therapeutics has the right to request appropriate modification to correct facts and to represent its opinions, or the opinions of the publication committee, if these differ with the proposed publication.